CLINICAL TRIAL: NCT06126393
Title: Study on the Prediction of Molecular Classification and Prognosis of Endometrial Cancer Using a Model Constructed by Magnetic Resonance Imaging Radiomics Combined With Pathomics
Brief Title: MRI Radiomics Combined With Pathomics on the Prediction of Molecular Classification and Prognosis of Endometrial Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Fujian Cancer Hospital (Other Government)
Collaborators: Fujian Provincial Hospital (Other); First Affiliated Hospital of Fujian Medical University (Other); Gutian Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHENJIAN1
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Endometrial Neoplasms
Keywords: Endometrial Neoplasms; machine learning; Radiomics; Pathomics; TCGA classification
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- POLE Mut: The POLE gene mutation detection was performed, and the mutation Changes were classified as POLE mutation.
  Interventions: Diagnostic Test: next generation sequencing AND Immunohistochemical examination
- dMMR: The mismatch repair (MMR) proteins were detected by immunohistochemistry, and the deletion of one or more proteins was classified as d-MMR subtype
  Interventions: Diagnostic Test: next generation sequencing AND Immunohistochemical examination
- P53abn: The expression of p53 was detected by immunohistochemistry. The abnormality of p53 protein expression (completely negative or diffusely strong positive in the nucleus) or expression location (cytoplasmic expression) was judged as p53abn, otherwise it was p53wt.
  Interventions: Diagnostic Test: next generation sequencing AND Immunohistochemical examination
- P53wt: The expression of p53 was detected by immunohistochemistry. The abnormality of p53 protein expression (completely negative or diffusely strong positive in the nucleus) or expression location (cytoplasmic expression) was judged as p53abn, otherwise it was p53wt.
  Interventions: Diagnostic Test: next generation sequencing AND Immunohistochemical examination

INTERVENTIONS:
Diagnostic Test: next generation sequencing AND Immunohistochemical examination — First, the mismatch repair (MMR) proteins were detected by immunohistochemistry, and the deletion of one or more proteins was classified as d-MMR subtype; Then the POLE gene mutation detection was performed, and the mutation Changes were classified as POLE mutation; Finally, p53 was detected by immunohistochemistry, and p53 mutant (p53 abn) and p53 wild-type (p53wt) were distinguished.
  Other Names: Magnetic resonance examination

SUMMARY:
Molecular typing provides accurate information for the diagnosis, treatment and prognosis prediction of endometrial cancer, which has important clinical significance. However, due to its high cost and complicated process, it is difficult to be widely used in clinical practice. Based on the artificial intelligence method, this study fused the characteristics of MRI radiomics and pathomics, combined with the clinical pathological information, built a model to predict the molecular typing and prognosis, analyzed the biological characteristics of endometrial cancer from the multi-scale level, guided the personalized and precise diagnosis and treatment, in order to improve the prognosis of patients.

DETAILED DESCRIPTION:
In this project, 150 cases of endometrial cancer were retrospectively collected, and 200 cases of endometrial cancer will be prospectively collected. All patients were pathologically confirmed and underwent Promise molecular typing. Before treatment, all patients completed abdominal MRI. Based on artificial intelligence technology, image features were extracted from magnetic resonance imaging, pathological features were extracted from pathological data, and clinical pathological data were collected at the same time. The treatment effect, recurrence and metastasis of patients were followed up, and the five-year survival rate and five-year progression free survival rate were calculated. It is proposed to focus on the following research:

1. Construction of molecular typing and prognosis prediction model of endometrial cancer based on magnetic resonance imaging Radiomics
2. Construction of molecular typing and prognosis prediction model of endometrial cancer based on pathomics.
3. Construction of a prediction model for molecular typing of endometrial cancer by integrating pathomics and radiomics.

ELIGIBILITY:
Inclusion Criteria:

* •Pathologically confirmed as endometrial malignant tumor with complete pathological H＆E stained sections;

  * Age ≥ 18 years and ≤ 80 years;
  * No other malignant cancers was found;
  * The complete immunohistochemical and second-generation sequencing results can be used for the molecular typing of ProMisE;
  * Magnetic resonance examination was performed within 2 weeks before treatment, and there was at least one measurable lesion according to RECIST 1.1 Criteria.

Exclusion Criteria:

* • The image quality is poor or the tumor is too small due to serious graphic artifact and degeneration, and the ROI cannot be accurately delineated;

  * Patients who received any antitumor therapy before surgery;
  * Diagnostic endometrial biopsy before MRI

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: 1. All patients were pathologically confirmed as endometrial malignant tumors, and molecular typing was performed.
  2. Patients with endometrial cancer who were admitted to Fujian cancer hospital from January 2020 to December 2023 were retrospectively collected. Meanwhile, from January 1, 2024, all consecutive patients with newly diagnosed endometrial cancer were enrolled and signed the informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Application of magnetic resonance imaging radiomics and pathomics to construct a model for predicting the molecular classification and prognosis of endometrial cancer | 2026-12-21
  The imaging and pathological features of endometrial cancer patients were extracted by artificial intelligence method. Combined with clinicopathological risk factors and survival time, an imaging nomogram was constructed by lasso regression method to predict the molecular classification and prognosis of endometrial cancer. ROC curve was used to evaluate the test efficiency of the model.

SECONDARY OUTCOMES:
Application of magnetic resonance imaging radiomics to construct a model for predicting the molecular classification and prognosis of endometrial cancer | 2026-12-21
  The imaging features of endometrial cancer patients were extracted by artificial intelligence method. Combined with clinicopathological risk factors and survival time, an imaging nomogram was constructed by lasso regression method to predict the molecular classification and prognosis of endometrial cancer. ROC curve was used to evaluate the test efficiency of the model.

OTHER OUTCOMES:
Application of pathomics to construct a model for predicting the molecular classification and prognosis of endometrial cancer | 2026-12-21
  The pathomics features of endometrial cancer patients were extracted by artificial intelligence method. Combined with clinicopathological risk factors and survival time, an imaging nomogram was constructed by lasso regression method to predict the molecular classification and prognosis of endometrial cancer. ROC curve was used to evaluate the test efficiency of the model.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Oncology School of Fujian Medical University, Fujian Cancer Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No
All relevant patient personal information and follow-up results of this study were saved by the principal investigator, and there was no plan to share them with other investigators

REFERENCES:
- [Result] Song XL, Luo HJ, Ren JL, Yin P, Liu Y, Niu J, Hong N. Multisequence magnetic resonance imaging-based radiomics models for the prediction of microsatellite instability in endometrial cancer. Radiol Med. 2023 Feb;128(2):242-251. doi: 10.1007/s11547-023-01590-0. Epub 2023 Jan 19. PMID 36656410
- [Result] Jamieson A, McAlpine JN. Molecular Profiling of Endometrial Cancer From TCGA to Clinical Practice. J Natl Compr Canc Netw. 2023 Feb;21(2):210-216. doi: 10.6004/jnccn.2022.7096. PMID 36791751
- [Result] Talhouk A, McConechy MK, Leung S, Li-Chang HH, Kwon JS, Melnyk N, Yang W, Senz J, Boyd N, Karnezis AN, Huntsman DG, Gilks CB, McAlpine JN. A clinically applicable molecular-based classification for endometrial cancers. Br J Cancer. 2015 Jul 14;113(2):299-310. doi: 10.1038/bjc.2015.190. Epub 2015 Jun 30. PMID 26172027
- [Result] Hou L, Zhou W, Ren J, Du X, Xin L, Zhao X, Cui Y, Zhang R. Radiomics Analysis of Multiparametric MRI for the Preoperative Prediction of Lymph Node Metastasis in Cervical Cancer. Front Oncol. 2020 Aug 20;10:1393. doi: 10.3389/fonc.2020.01393. eCollection 2020. PMID 32974143
- [Result] Lefebvre TL, Ueno Y, Dohan A, Chatterjee A, Vallieres M, Winter-Reinhold E, Saif S, Levesque IR, Zeng XZ, Forghani R, Seuntjens J, Soyer P, Savadjiev P, Reinhold C. Development and Validation of Multiparametric MRI-based Radiomics Models for Preoperative Risk Stratification of Endometrial Cancer. Radiology. 2022 Nov;305(2):375-386. doi: 10.1148/radiol.212873. Epub 2022 Jul 12. PMID 35819326
- [Result] Crosbie EJ, Kitson SJ, McAlpine JN, Mukhopadhyay A, Powell ME, Singh N. Endometrial cancer. Lancet. 2022 Apr 9;399(10333):1412-1428. doi: 10.1016/S0140-6736(22)00323-3. PMID 35397864